CLINICAL TRIAL: NCT06459557
Title: Management of Pediatric Distal Radius Fractures : Conservative Treatment Versus Surgical Reduction - a Randomized Controlled Trial
Brief Title: Management of Pediatric Distal Radius Fractures : Conservative Treatment Versus Surgical Reduction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Hasan Mohamed, resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: casting of distal radius
Record Dates: First submitted 2024-05-12; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Fracture, Radius
MeSH Terms: conditions — Radius Fractures | interventions — POLR1G protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservative treatment of displaced pediatric distal radius fractures (Active Comparator): children in this group with displaced distal radius fractures would be managed by a cast in the emergency room without anatomically reducing the fracture under general anesthesia in the operating room
  Interventions: Procedure: cast
- surgical reduction of displaced distal radius fractures (Active Comparator): children in this group with displaced distal radius fractures would be managed by being anatomically reducing the fracture in the operating room under general anesthesia
  Interventions: Procedure: surgical reduction

INTERVENTIONS:
Procedure: cast — children with displaced distal radius fractures would be managed by a cast in the emergency room
  Arms: conservative treatment of displaced pediatric distal radius fractures
Procedure: surgical reduction — anatomical reduction of pediatric displaced distal radius fractures under general anesthesia in the operating room
  Arms: surgical reduction of displaced distal radius fractures

SUMMARY:
To compare functional and radiological assessment between two groups of children with displaced distal radius fractures : those who will receive surgical reduction and those who will not.

DETAILED DESCRIPTION:
Distal radius fractures are the most frequent fractures seen in pediatric population accounting for about 20-30% of all fractures in children , for the non-displaced pediatric distal radius fractures , it is agreed widely to be just managed by an immobilization cast in the emergency department . However when it comes to the displaced fractures , Different centers have different options of management , mostly including either the surgical anatomical reduction under general anesthesia then casting with or without using other fixation method which is mostly k-wires , or the other option includes only casting in the emergency department without trial of reduction or just a trial of realignment under sedating agent , this second option depends on the unique phenomenon of remodeling in the pediatric fractures , as Unlike adults, in growing children, remodeling can restore the alignment of the displaced fractures to a certain extent, making anatomical reduction less essential , specially when it comes to distal radius as The distal radial and ulnar physes are responsible for about 80% of forearm length and for 40% of upper limb length that making their remodeling potential can approach upto 100% . depending on that the question was that if the fracture will be fully remodeled with no functional or range of motion disturbance on the conservative option so what the essentiality of the surgical option can be . along with exposing the child to the dangers of general anesthesia , the minor complications that can occur with k wires (as neuropraxia , pin tract infection or migration of the k wire) , emotional and financial load . in a cost analysis for different options of treatment in displaced pediatric distal radius fractures , the cost of surgical option exceeds the conservative one by multiple times . According to that a lot of the current literature have suggested to consider conservative treatment of pediatric displaced distal radius fractures to be the gold standard and fundamental option of treatment . In this study the investigators question the effectiveness of conservative treatment to displaced pediatric distal radius fractures (casting in the emergency department) in comparison to the surgical anatomical reduction in matters of functional and radiological parameters .

ELIGIBILITY:
Inclusion Criteria:

* All children aged 3 to 10 years
* both genders
* patients presenting with displaced distal radius fractures

Exclusion Criteria:

* intra articular fractures
* Greenstick and buckle fractures
* fractures with more than 1 week duration
* non displaced fractures
* Salter Harris fractures
* open fractures
* fractures with neurovascular bundle injury
* poly trauma patients
* patients with pathological bone diseases as Osteogenesis Imperfecta or CP (cerebral palsy) .
* Galeazzi fractures

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
mean difference of Modifed the Disabilities of the Arm, Shoulder and Hand (m-DASH) score between the two groups | 12 months
  functional assessment at 1.5 , 3 , 6 and 12 months posttrauma using the Modifed the Disabilities of the Arm, Shoulder and Hand (m-DASH) score as (50/50) (100%) is considered the maximum value which is the best outcome and (10/50) (0%) is considered the minimum value which is the worst outcome

SECONDARY OUTCOMES:
Comparing palmar tilt angle between the 2 groups . | 12 months
  radiological assessment poattraumatic at 1.5 , 3 , 6 ,12 months for lateral view of wrist joint for the 2 groups comparing palmar tilt angle which is the angle formed by a line drawn perpendicular to the axis of the radial shaft, and a line that passes through the tips of the dorsal and volar rims (i.e. along the radius articular surface)
Comparing radial inclination between the 2 groups | 12 months
  radiological assessment posttraumatic at 1.5 , 3 , 6 ,12 months for anterioposterior view of wrist joint for the 2 groups comparing radial inclination which is the angle between a line drawn perpendicular to the long axis of the radius along the articular surface of the distal radius and a line drawn down from the tip of the radial styloid
Comparing radius length between the 2 groups | 12 months
  radiological assessment posttraumatic at 1.5 , 3 , 6 ,12 months for anterioposterior view of wrist joint for the 2 groups comparing radius length which is the distance between two lines drawn perpendicular to the long axis of the radius on the AP projection from the apex of the radial styloid and level of the ulnar aspect of the articular surface

REFERENCES:
- [Background] Akar D, Koroglu C, Erkus S, Turgut A, Kalenderer O. Conservative Follow-up of Severely Displaced Distal Radial Metaphyseal Fractures in Children. Cureus. 2018 Sep 5;10(9):e3259. doi: 10.7759/cureus.3259. PMID 30430048
- [Background] Shah AS, Guzek RH, Miller ML, Willey MC, Mahan ST, Bae DS; Pediatric Distal Radius Fracture (PDRF) Study Group. Descriptive Epidemiology of Isolated Distal Radius Fractures in Children: Results From a Prospective Multicenter Registry. J Pediatr Orthop. 2023 Jan 1;43(1):e1-e8. doi: 10.1097/BPO.0000000000002288. Epub 2022 Oct 26. PMID 36299238
- [Background] Hove LM, Brudvik C. Displaced paediatric fractures of the distal radius. Arch Orthop Trauma Surg. 2008 Jan;128(1):55-60. doi: 10.1007/s00402-007-0473-x. Epub 2007 Oct 17. PMID 17940779
- [Background] Sengab A, Krijnen P, Schipper IB. Displaced distal radius fractures in children, cast alone vs additional K-wire fixation: a meta-analysis. Eur J Trauma Emerg Surg. 2019 Dec;45(6):1003-1011. doi: 10.1007/s00068-018-1011-y. Epub 2018 Oct 1. PMID 30276723
- [Background] Marinelli M, Massetti D, Facco G, Falcioni D, Coppa V, Maestri V, Gigante A. Remodeling of distal radius fractures in children: preliminary retrospective cost/analysis in level II pediatric trauma center. Acta Biomed. 2021 Nov 3;92(5):e2021390. doi: 10.23750/abm.v92i5.11971. PMID 34738560
- [Background] Naik P. Remodelling in Children's Fractures and Limits of Acceptability. Indian J Orthop. 2021 Mar 10;55(3):549-559. doi: 10.1007/s43465-020-00320-2. eCollection 2021 Jun. PMID 33995859
- [Background] Orland KJ, Boissonneault A, Schwartz AM, Goel R, Bruce RW Jr, Fletcher ND. Resource Utilization for Patients With Distal Radius Fractures in a Pediatric Emergency Department. JAMA Netw Open. 2020 Feb 5;3(2):e1921202. doi: 10.1001/jamanetworkopen.2019.21202. PMID 32058553
- [Background] Colovic H, Stankovic I, Dimitrijevic L, Zivkovic V, Nikolic D. The value of modified DASH questionnaire for evaluation of elbow function after supracondylar fractures in children. Vojnosanit Pregl. 2008 Jan;65(1):27-32. doi: 10.2298/vsp0801027c. PMID 18368935